CLINICAL TRIAL: NCT00483041
Title: A Phase2A, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Effect of a Single-Dose Intravenous Administration of MEDI-528, A Humanized Anti-Interleukin-9 Monoclonal Antibody, on Allergen-Induced Interleukin-9 Levels in Bronchoalveolar Lavage Fluid in Adults With Atopic Asthma
Brief Title: A Study to Evaluate the Effect of a Single-Dose Intravenous Administration of MEDI-528
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study is replaced by MI-CP198 per CPM.
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MI-CP139
Record Dates: First submitted 2007-06-04; First posted 2007-06-06 (Estimated); Results first posted 2014-03-07 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — enokizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- MEDI528 9 mg/kg (Experimental): MEDI-528 at a dose of 9 mg/kg administered as a single intravenous infusion
  Interventions: Biological: MEDI528 9 mg/kg
- PLACEBO (Placebo Comparator): Placebo administered as a single intravenous infusion
  Interventions: Other: PLACEBO

INTERVENTIONS:
Other: PLACEBO — Placebo administered as a single intravenous infusion
  Arms: PLACEBO
Biological: MEDI528 9 mg/kg — MEDI-528 at a dose of 9 mg/kg administered as a single intravenous infusion
  Arms: MEDI528 9 mg/kg

SUMMARY:
To evaluate the effect of MEDI-528 in adults with atopic asthma.

DETAILED DESCRIPTION:
To evaluate the effect of MEDI-528 on the change in biologically active IL-9 levels in BAL fluid following segmental allergen challenge in adults with atopic asthma.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults, age 18 through 50 years of age at time of screening;
* Written informed consent obtained from the patient prior to receipt of any study medication or beginning any study procedures;
* Previously documented diagnosis of asthma based on episodic symptoms of airflow obstruction such as wheezing or chest tightness, with alternative diagnoses (eg, chronic obstructive pulmonary disease) ruled out;
* Forced expiratory volume in one second (FEV1) ≥ 70% of predicted value;
* A positive skin prick or intradermal test to cat allergen extract, short ragweed allergen extract, or dust mite allergen extracts. A positive skin test is defined as the indurations of skin test wheal being at least 2 mm greater in diameter than that of the indurations of the control skin wheal;
* History of asthmatic symptoms upon exposure to at least one of the allergens (cat allergen extract, short ragweed allergen extract, or dust mite allergen extracts) that induces a positive skin prick test;
* AHR on methacholine inhalation challenge test, with PC20 ≤ 8 mg/mL (Crapo, 2000);
* No significant changes in regular asthma medications and no acute asthma exacerbations requiring oral corticosteroids or doubling of ICS dosage, hospitalization, emergency room visits, or unscheduled health care provider visits for asthma for at least 6 weeks prior to screening and up through the time of study drug administration;
* No history of intubation or admission to an intensive care unit for asthma;
* Sexually active women, unless surgically sterile or at least 1 year post-menopausal, must have used an effective method of avoiding pregnancy (including oral or implanted contraceptives, intrauterine device, female condom, diaphragm with spermicide, cervical cap, abstinence, use of a condom by the sexual partner or sterile sexual partner) for 21 days prior to the study drug administration on Study Day 0, and must agree to continue using such precautions through Study Day 126. Cessation of birth control after this point should be discussed with a responsible physician. Sexually active men, unless surgically sterile, must likewise use an effective method of birth control (condom) and must agree to continue using such precautions through Study Day 126;
* Able to follow study procedures including the ability to provide spirometry readings that meet American Thoracic Society (ATS)/European Respiratory Society (ERS) standards (Miller, 2005);
* Ability to complete the study period, including follow-up period, of up to 126 days; and
* Willing to forego other forms of experimental treatment and study procedures during study.

Exclusion Criteria:

* Receipt of MEDI-528 in any previous clinical study;
* History of allergy or reaction to any component of the study drug formulation or other medications, such as topical lidocaine, administered during bronchoscopy;
* Lung disease other than allergic asthma (eg, chronic bronchitis);
* FEV1 < 70% of predicted values;
* Use of systemic immunosuppressive drugs including systemic corticosteroids (topical corticosteroids are permitted), ICS at doses > 800 μg/day budesonide or equivalent, long-acting β2 agonists (eg, salmeterol), leukotriene antagonists, cromolyn sodium, nedocromil sodium, theophylline, omalizumab, or any other medication for asthma except short-acting β2 agonist (as needed) within the 4 weeks prior to screening up through administration of study drug;
* Current use of any β-adrenergic antagonist (eg, propranolol);
* Any disease or illness, other than asthma, that may require the use of systemic corticosteroids during the study period;
* Upper or lower respiratory tract infections within 8 weeks before screening;
* Acute illnesses or evidence of clinically significant active infection, such as fever ≥ 38.0°C (100.5°F) at screening and through the time of the study drug administration on Study Day 0;
* Current allergy vaccination therapy (desensitization immunotherapy) with less than 3 months of stable maintenance doses prior to the baseline segmental allergen challenge. The allergy vaccination must not include desensitization to the allergen that will be used in the segmental allergen challenge;
* Receipt of any investigational drug therapy within 30 days or any biologic(s) within 5 half-lives of the agent prior to study drug administration through Study Day 126;
* Receipt of any therapy with a leukocyte-depleting agent (eg, rituximab, alemtuzumab) unless recovery in white cell count has been documented before screening;
* Pregnancy (sexually active females must have negative serum and urine pregnancy tests at screening and a negative urine pregnancy test prior to study drug administration on Study Day 0);
* Is a nursing mother at the time of screening;
* Evidence of infection with hepatitis B or C virus, or HIV-1 or HIV-2, or active infection with hepatitis A;
* History of significant systemic disease (eg, cancer, infection, hematological, renal, hepatic, coronary artery disease or other cardiovascular disease, endocrinologic, neurologic, rheumatologic, or gastrointestinal disease);
* History of cancer other than basal cell carcinoma or cervical carcinoma-in-situ treated with apparently successful curative therapy (remission for ≥ 1 year prior to screening);
* History of primary immunodeficiency;
* History of pancreatitis or currently active gastroduodenal ulcer;
* History of coagulation disorders or abnormal PT and PTT test results at screening;
* History of life-long urinary retention;
* History of use of tobacco products of more than one cigarette per month or equivalent within 1 year prior to screening or history of smoking of ≥ 10 pack-years;
* History of anaphylaxis;
* Elective surgery planned from the time of screening through Study Day 126;
* Clinically significant abnormalities (other than asthma) upon physical examination prior to study drug administration on Study Day 0;
* Clinically significant abnormality, as determined by the investigator, on 12-lead ECG or chest radiograph at the time of screening;
* At the time of screening, any of the following: hemoglobin, total white blood cell count (WBC), platelet count, sodium (Na), potassium (K), chloride (Cl), or carbon dioxide (CO2)out of the normal range; aspartate transaminase (AST), alanine transaminase (ALT), blood urea nitrogen (BUN), amylase, lipase, or serum creatinine above the upper limits of normal (ULN); or other abnormal laboratory values in the screening panel that are judged by the principal investigator to be clinically significant; or
* No detectable levels of IL-9 in the Baseline Visit 2' BAL sample, or any finding upon physical examination or history of any disease that, in the opinion of the principal investigator or medical monitor, may compromise the safety of the patient in the study or confound the analysis of the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2007-07; Primary Completion 2008-10 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Parker, M.D., Study Director — MedImmune LLC
Locations (4):
- United States (4):
  - Brigham & Women's Hospital Asthma Research, Boston, Massachusetts
  - Washington Univeristy School of Medicine, Division of Pulmonary and Critical Care Medicine, St Louis, Missouri
  - Wake Forest University, Baptist Medicial Center, Winston-Salem, North Carolina
  - University of Wisconsin, Section of Allergy, Pulmonary & Critical Care, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 11 adult participants participated in the study between 19Jul2007 and 15Oct2008 at 2 sites in the United States of America.
Pre-assignment Details: Treatment assignments were determined using a block randomization procedure with a 1:1 ratio through an interactive voice response system. Only participants who had detectable levels of interleukin-9 in the Baseline Visit 2' bronchioalveolar lavage sample will be randomized.
Groups:
- PLACEBO: Placebo administered as a single intravenous dose
- MEDI528 9 mg: MEDI-528 at a dose of 9 mg/kg administered as a single intravenous infusion
Period: Overall Study
Arm/Group | PLACEBO | MEDI528 9 mg
Started | 5 | 6
Completed | 5 | 5
Not Completed | 0 | 1
Not completed — ABNORMAL LAB DATA AT SCREENING | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PLACEBO | MEDI528 9 mg | Total
Number analyzed (Participants) | 5 | 6 | 11
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.2 (7.8) | 22.3 (2.7) | 25.5 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 2 | 5 | 7

OUTCOME MEASURES:

1. Primary Outcome: Listing of Total Interleukin-9 (IL-9) Counts by Enzyme-linked Immunosorbent Assay in Bronchoalveolar Lavage Fluid (BAL)
Description: The response of biologically active IL-9 in BAL fluid to the segmental allergen challenge, 1-2 days after the applying the allergen, prior to and 2 weeks after investigational product administration.
Time Frame: Baseline (2 to 4 weeks prior to Day 0) and Day 15
Population: All subjects who were randomized (n=11), received at least one dose of investigational product (MEDI-528 or placebo; n=10), and completed the 2-day BAL and segmental allergen challenge procedures at baseline (2-4 weeks prior to Day 0) and on Days 14 and 15 (n=2; 1 subject in each treatment group).
Measure: Number; unit: Picograms per milliliter
Arm/Group | PLACEBO | MEDI528 9 mg/kg
Number analyzed (Participants) | 1 | 1
Picograms per milliliter
  Baseline | 8.31 (0) | 4.04 (0)
  Day 15 | 40.05 | 43.01

2. Secondary Outcome: Incidence of Adverse Events
Description: Number of participants experiencing adverse events (includes both adverse events and serious adverse events)
Time Frame: Days 0 - 126
Population: All participants who were randomized (n=11) and received at least one dose of investigational product (MEDI-528 or placebo; n=10).
Measure: Number; unit: Participants
Arm/Group | PLACEBO | MEDI528 9 mg/kg
Number analyzed (Participants) | 5 | 5
Participants | 5 | 5

3. Secondary Outcome: Incidence of Serious Adverse Events
Description: Number of participants experiencing serious adverse events
Time Frame: Days 0 - 126
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | PLACEBO | MEDI528 9 mg/kg
Number analyzed (Participants) | 5 | 5
Participants | 0 | 0

4. Secondary Outcome: Incidence of Anti-drug Antibodies (ADA) to MEDI-528
Description: Number of participants with ADA to MEDI-528
Time Frame: Days 0, 28, 56, 84, and 126
Population: All participants who were randomized (n=11) and received at least one dose of investigational product (MEDI-528 or placebo; n=10). One subject in the 9 mg/kg group had no sample collected on Day 126.
Measure: Number; unit: Participants
Arm/Group | PLACEBO | MEDI528 9 mg/kg
Number analyzed (Participants) | 5 | 5
Participants | 0 | 0

5. Secondary Outcome: Time to Peak Concentration (Tmax)
Description: Tmax of MEDI-528
Time Frame: Days 0, 1, 7, 14, 15, 28, 56, 84, and 126
Population: All participants who were randomized (n=11), received MEDI-528 (n=5), and had pharmacokinetic samples for analysis (n=4)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day
Arm/Group | PLACEBO | MEDI528 9 mg/kg
Number analyzed (Participants) | 0 | 4
Day |  | 0.040 (88.4)

6. Secondary Outcome: Peak Concentration (Cmax)
Description: Cmax of MEDI-528
Time Frame: Days 0, 1, 7, 14, 15, 28, 56, 84, and 126
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | PLACEBO | MEDI528 9 mg/kg
Number analyzed (Participants) | 0 | 4
Microgram per milliliter |  | 210.634 (23.9)

7. Secondary Outcome: Area Under the Concentration Curve From Time Zero to Last Measurable Concentration [AUC(0-t)]
Description: AUC(0-t) of MEDI-528
Time Frame: Days 0, 1, 7, 14, 15, 28, 56, 84, and 126
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram times day per milliliter
Arm/Group | PLACEBO | MEDI528 9 mg/kg
Number analyzed (Participants) | 0 | 4
Microgram times day per milliliter |  | 4347.489 (24.1)

8. Secondary Outcome: Area Under the Concentration Curve From Time Zero to Infinity [AUC(0-infinity)]
Description: AUC(0-infinity) of MEDI-528
Time Frame: Days 0, 1, 7, 14, 15, 28, 56, 84, and 126
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram times day per milliliter
Arm/Group | PLACEBO | MEDI528 9 mg/kg
Number analyzed (Participants) | 0 | 4
Microgram times day per milliliter |  | 4845.344 (17.8)

9. Secondary Outcome: Percent of Total Area Under the Concentration Curve Extrapolated From Last Measurable Time to Infinity [AUC(Ext)]
Description: AUC(ext) of MEDI-528
Time Frame: Days 0, 1, 7, 14, 15, 28, 56, 84, and 126
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of Total Area
Arm/Group | PLACEBO | MEDI528 9 mg/kg
Number analyzed (Participants) | 0 | 4
Percentage of Total Area |  | 8.283 (78.8)

10. Secondary Outcome: Clearance (CL)
Description: CL of MEDI-528
Time Frame: Days 0, 1, 7, 14, 15, 28, 56, 84, and 126
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milliliters per day
Arm/Group | PLACEBO | MEDI528 9 mg/kg
Number analyzed (Participants) | 0 | 4
Milliliters per day |  | 167.702 (2.7)

11. Secondary Outcome: Terminal Half-life (T1/2)
Description: T1/2 of MEDI-528
Time Frame: Days 0, 1, 7, 14, 15, 28, 56, 84, and 126
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Day
Arm/Group | PLACEBO | MEDI528 9 mg/kg
Number analyzed (Participants) | 0 | 4
Day |  | 32.134 (3.6)

12. Secondary Outcome: Volume at Steady State (Vss)
Description: Vss of MEDI-528
Time Frame: Days 0, 1, 7, 14, 15, 28, 56, 84, and 126
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milliliter
Arm/Group | PLACEBO | MEDI528 9 mg/kg
Number analyzed (Participants) | 0 | 4
Milliliter |  | 7354.025 (5.6)

13. Secondary Outcome: Volume at Distribution (Vz)
Description: Vz of MEDI-528
Time Frame: Days 0, 1, 7, 14, 15, 28, 56, 84, and 126
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milliliter
Arm/Group | PLACEBO | MEDI528 9 mg/kg
Number analyzed (Participants) | 0 | 4
Milliliter |  | 7772.894 (3.5)

ADVERSE EVENTS:
Arm/Group | PLACEBO | MEDI528 9 mg
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 5/5 | 5/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PLACEBO (N=5) | MEDI528 9 mg (N=5)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 2 (2)
Allergy to animal (Immune system disorders) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2)
Post procedural complication (Injury, poisoning and procedural complications) | 4 (15) | 5 (7)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Post procedural swelling (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural headache (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Breath sounds abnormal (Investigations) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Migraine with aura (Nervous system disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Nasal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome. The PIs also agree for data to be presented first as a joint, multi-center publication.